CLINICAL TRIAL: NCT02504632
Title: Study of Platelet Activation by Severe Aortic Stenosis and Its Correction by Transcatheter Aortic Valve Implantation (TAVI) Platelet Activation in TAVI
Brief Title: Study of Platelet Activation by Severe Aortic Stenosis and Its Correction by Transcatheter Aortic Valve Implantation
Acronym: TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14 7078 03
Record Dates: First submitted 2015-07-17; First posted 2015-07-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Aortic Stenosis
Keywords: platelet activation; transcatheter aortic valve implantation
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test group (Experimental): Patient with severe, symptomatic AS (Aortic valve area < 0,6 cm2/m2 SC), deemed, after multidisciplinary heart team evaluation, contra-indicated or at high risk for surgery and suitable for TF TAVI with a MCV prosthesis.
  Interventions: Other: test
- control group (Other): Patient with stable coronary artery disease, unscathed of AS Patient under aspirin treatment (75-160 mg/d for at least one week)
  Interventions: Other: control group

INTERVENTIONS:
Other: test — Peripheral venous citrated blood will be collected just before and 10-15 min after the implantation of the valve. Samples will be obtained after starting the infusion of contrast media. In peripheral venous blood before 24 h and after the procedure and at hospital discharge, 4-6 days when the usual transient thrombocytopenia after TAVI has recovered.
  The results will be used to analyse the kinetics of haematological changes in peripheral blood following aortic valve replacement.
  Platelet activation will be monitored by flow cytometry to assess the expression of specific membrane markers and the phosphorylation of signalling proteins, as well as the formation of platelet/monocyte aggregates.
  Arms: test group
Other: control group — In this group, only one sample (2 tubes filled with 4.5 ml, i.e. 9ml) will be obtained in venous peripheral blood to establish reference values in age-matched, aspirin-treated, atherosclerotic population.
  Arms: control group

SUMMARY:
Study of platelet activation by severe aortic stenosis and its correction by Transcatheter Aortic Valve Implantation (TAVI)

DETAILED DESCRIPTION:
* Background: TAVI has emerged as an alternative to surgical aortic valve replacement for patients with severe, symptomatic aortic stenosis (AS) and is expanding worldwide with more than 50,000 patients treated to date.
* Purpose Changes in haemostasis, particularly in platelet activation or reactivity before, during and after TAVI have never been studied. Valve replacement is known to alleviate von Willebrand factor abnormalities associated with AS. A potential improvement of platelet function could also occur after TAVI. Indeed, circulating platelets may be desensitized and under-reactive due to multiple passages through the stenotic valve and could recover normal reactivity after TAVI. Besides, TAVI presents a risk of major ischemic complications. The investigators can hypothesize the involvement of high reactive platelets in peri-procedural thrombotic or ischemic events. This study of the platelet activation kinetics will be performed by comparing several specific markers before and at various times after valve implantation.
* Primary outcome To evaluate the kinetics of platelet activation before and at various times after valve implantation, by comparing several specific markers in peripheral venous blood samples before (day 0) and at days 1 and 5±1 after the procedure.
* Study design and number of subjects: This is a prospective, monocentric, study. The test group includes up to 15 patients treated by transfemoral TAVI using a MedTronic CoreValve (MCV) prosthesis. Platelet activation will be studied before and after the procedure and compared to a reference established with an age-matched, aspirin-treated, atherosclerotic population (30 patients in the control group).
* Eligibility criteria:

  * inclusion criteria: test group: patients with severe aortic stenosis and transfemoral TAVI with MCV aspirin treatment . Control group: age-matched patients with stable coronary artery disease treated by aspirin but without aortic stenosis.
  * exclusion criteria: recent (1 month) acute coronary syndrome; treatment by anti platelet agents other than aspirin
* Procedures: Specific platelet activation markers, circulating platelet/monocytes aggregates, platelet reactivity and vWF will be assessed in peripheral venous blood before, 1 and 5 days after TAVI and in ascending aorta during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Test group

  * Severe symptomatic AS (Aortic valve area < 0,6 cm2/m2 SC), deemed, after multidisciplinary heart team evaluation, contra-indicated or at high risk for surgery and suitable for TF TAVI with a MCV prosthesis.
  * Aspirin treatment (75-160 mg/d for at least one week)
* Control group

  * Stable coronary artery disease, unscathed of AS
  * Aspirin treatment (75-160 mg/d for at least one week)

Exclusion Criteria:

* Test group:

  * Acute coronary syndrome 1 month before inclusion
  * Any co-morbidity limiting life-expectancy < 1 year
  * Terminal chronic kidney disease requiring hemodialysis thrombocytopenia <100 G/L, anemia (Hb < 10 g/dl)
  * Treatment by another antiplatelet agent within 10 days before the procedure
* Control group:

  * Acute coronary syndrome 1 month before inclusion
  * Any co-morbidity limiting life-expectancy < 1 year
  * Terminal chronic kidney disease requiring hemodialysis
  * Thrombocytopenia <100 G/L
  * Treatment by another antiplatelet agent within 10 days before the procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the change of kinetics of platelet activation | 1 min before TAVI and at days 1after TAVI
  Evaluate the kinetics of platelet activation before and at various times after valve implantation, by comparing several specific markers in peripheral venous blood samples before (day 0) and at day 1 after the procedure using flow cytometry (FACS).
the change of kinetics of platelet activation | 1 min before TAVI and 5±1 after TAVI
  Evaluate the kinetics of platelet activation before and at various times after valve implantation, by comparing several specific markers in peripheral venous blood samples before (day 0) and at 5±1 days after the procedure using flow cytometry (FACS).

SECONDARY OUTCOMES:
Changes of platelet activation | 1 min before and 10 min after TAVI
  platelet activation in aortic blood downstream of the stenotic valve before and 10 min after TAVI,
Changes of platelet activity | 1 min before and day 1 after TAVI
  platelet reactivity to selected agonists in peripheral venous blood samples before and at days 1 and 5±1. Measure of platelet/monocytes aggregates by flow cytometry approaches. Measure of plasma serotonin and soluble GPIV by an by an ELISA technique
Changes of platelet activity | 1 min before and day 5 after TAVI
  platelet reactivity to selected agonists in peripheral venous blood samples before and at days 1 and 5±1,
changes in von Willebrand factor | 1 min before and day 1 and 5 after TAVI
  changes in von Willebrand factor in peripheral blood samples The activity and level of vWF antigen will be measured by immunotubidimetric methods

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SIE, MD PhD, Study Chair — University Hospital, Toulouse
Locations (1):
- CHU TOULOUSE-Hôpital Rangueil, Toulouse, France